CLINICAL TRIAL: NCT05314530
Title: Validation of the ReTA-model: Rehabilitation Trail for Workers on Long-term Sick Leave in the Healthcare
Brief Title: The ReTA-model: Rehabilitation Trail for Workers on Long-term Sick Leave in the Healthcare Sector
Acronym: ReTA-model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emma Hagqvist, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReTA-model
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Burnout
Keywords: Healthcare; Burnout; Stress; Return to work; Intervention
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Will receive a rehabilitation intervention
  Interventions: Behavioral: ReTA-model
- Controll (Active Comparator): Will receive conventional rehabilitation
  Interventions: Behavioral: ReTA-model

INTERVENTIONS:
Behavioral: ReTA-model — Validating the rehabilitation model ReTA

SUMMARY:
The ReTA-model is a rehabilitation model for return to work after long-term sickness absence (LTSA) due to stress or burnout. The ReTA-model will be validated in this trial among nurses and physicians currently in LTSA. The ReTA-model includes a three-week treatment with exercise, individual and collegial talks with psychology and lecturing. The control group will receive conventional rehabilitation from regular care.

DETAILED DESCRIPTION:
The ReTA-model is a rehabilitation model for return to work after long-term sickness absence (LTSA) due to stress or burnout. The ReTA-model will be validated in this trial among nurses and physicians currently in LTSA. The ReTA-model includes a three-week treatment with exercise, individual and collegial talks with psychology and lecturing. The control group will receive conventional rehabilitation from regular care.

ELIGIBILITY:
Inclusion Criteria:

* currently on sick leave for burnout
* employed in the Swedish healthcare services as a nurse or as a physician

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Return to work | 12 months
  At work part or full-time compare to no return to work
Karolinska Exhaustion Disorder Scale KEDS | 12 months
  Decreased points in the KEDS scale 1-19, qith higher scores reflecting greater exhaustion severity.
Symptom Checklist - 6 | 12 months
  Decreased points on the SCL-6 scale, with a higher number reflecting depression.
Montgomery Åsberg Depression Rating Scale | 12 months
  Decreased points in the MADRAS scale with score ranging from 0 to 60, with higher scores reflecting greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hagqvist, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Outside U.S. and Canada, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thunqvist E, Nygren A, Lofman B, Parker D, Brulin E. Assessing the Effect of a Rehabilitation Intervention on Exhaustion Disorders, Depression, and Return to Work: A Randomized Controlled Trial. J Occup Rehabil. 2025 Dec 13. doi: 10.1007/s10926-025-10350-y. Online ahead of print. PMID 41389236